CLINICAL TRIAL: NCT06520605
Title: Cytomegalovirus Reactivation in Non-immunosuppressed Patients Requiring Prolong Mechanical Ventilation
Brief Title: Cytomegalovirus Reactivation in ICU Patients Requiring Prolong Mechanical Ventilation
Status: Recruiting | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2024-122-DM-138
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Ventilation
Keywords: Critical Illnesses; Virus Activation; Cytomegalovirus
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cytomegalovirus (CMV) is a latent infection virus that is widespread in the population. CMV may reactivate under certain circumstances, and its hazardous nature has been proven, especially in immunosuppressed patients. However in recent years, some studies have found that CMV reactivation also exists in apparently immunocompetent patients during their critical illness. In these non-immunosuppressed patients, the presence of sepsis and its immunomodulatory effects may lead to reactivation of dormant viral infections. Studies found the incidence of CMV reactivation in up to one-fourth to half of these non-immunosuppressed patients during their critical illness.

These studies also documented significantly higher length of ICU stay and mortality in critically ill patients with CMV reactivation. CMV reactivation has also been studied in specific critically ill cohorts, exhibiting there impact on mortality. David S Y Yong et al studied the effect of CMV reactivation on mortality in immunocompetent acute respiratory distress syndrome (ARDS) patients. In a recent study, it was found that among cohort of non-immunosuppressed patients with acute respiratory distress syndrome (ARDS), CMV reactivation occurred in 27 % of patients which was associated with overall increased ICU mortality. In another study among septic shock cohort (329 patients), herpesvirus reactivations were documented in 68% patients without prior immunodeficiency and concluded that reactivations could be independently associated with mortality.

However currently, no study is available investigating the CMV reactivation and it's kinetics during critical illness in non immunocompetent patients requiring prolonged mechanical ventilation. In this planned observational study, we aim to find out the prevalence of Cytomegalovirus (CMV) reactivation, viral load and it's association with the severity of illness in non immunosuppressed ICU patients requiring prolong mechanical ventilation.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is a latent infection virus that is widespread in the population. CMV may reactivate under certain circumstances, and its hazardous nature has been proven, especially in immunosuppressed patients. However, several studies have found that CMV reactivation also exists in immunocompetent patients with a critical illness. Among those patients, the incidence of CMV reactivation, which is more than 30%, is associated with increased duration of hospital stay, and higher mortality.

Traditionally, critically ill patients have been considered immunocompetent but the presence of sepsis and its immunomodulatory effects may lead to reactivation of dormant viral infections. Sepsis due to its immunomodulatory effects may lead to reactivation of CMV due to the release of pro-inflammatory cytokines such as TNF-alpha and IL-1beta which has the ability to activate several transcription factors contributing in the CMV reactivation. Clari et al showed that CMV infection in critically ill patients was consistently associated with undetectable IFN-γ T cell responses within the first 2 days of admission to the ICU, and that viral load was inversely related to IFN-γ T cell responses. Similar results were also found by Venet et al that septic patients display immune system paralysis, reduced Th1 cell function, increased IL-10 production (anti-inflammatory), global lymphopenia affecting natural killer cells (NK) quantitatively and qualitatively related to their interferon production.

Studies have documented significantly higher organ failure rates and mortality in critically ill patients with CMV reactivation. Phillips Lachance et al performed a systematic review to investigate the association between CMV reactivation and clinical outcomes in immunocompetent critically ill patients. In this review, twenty-two studies were included. CMV reactivation was associated with increased ICU mortality, overall mortality, duration of mechanical ventilation, nosocomial infections, ICU length of stay. CMV reactivation has also been studied in specific critically ill cohorts, exhibiting there impact on mortality. David S Y Yong et al studied the effect of CMV reactivation on mortality in immunocompetent acute respiratory distress syndrome (ARDS) patients. Of 399 ARDS patients, 68 % were CMV seropositive and reactivation occurred in 27 % of them which was associated with overall increased ICU mortality. In another study among septic shock cohort (329 patients), herpesvirus reactivations were documented in 68% patients without prior immunodeficiency and concluded that reactivations could be independently associated with mortality.

However, currently no study is currently available investigating the CMV reactivation and it's kinetics during critical illness in non-immunosuppressed patients requiring prolonged mechanical ventilation. In this planned observational study, the investigators aimed to find out the prevalence of CMV reactivation, viral load and it's association with the severity of illness in non-immunosuppressed ICU patients requiring prolong mechanical ventilation.

All adult ICU patients requiring prolong mechanical ventilation will be considered for inclusion and will be screened for the presence of Anti CMV IgG antibodies in blood. If patient is IgG seropositive and meets inclusion/ exclusion criteria, then they will be included in study and will be followed up for CMV reactivation during their ICU stay (on weekly basis till maximum 28-days after the initiation of mechanical ventilation). In patients who had CMV reactivation, viral load kinetics will be further followed up on weekly basis for the next 3 weeks or ICU discharged (whichever comes first). Blood samples will be collected in all; while tracheal aspirate sample will be collected in whom who had an artificial airway.

ELIGIBILITY:
Inclusion Criteria:

* All adult ICU patients requiring prolonged mechanically ventilation (at least 7 days of supportive ventilation) and the presence of CMV seropositivity (Anti CMV IgG antibodies) will be considered for inclusion

Exclusion Criteria:

* Age <18 years
* Use of anti viral agent within last 7 days
* Duration of mechanical ventilation more than 14 days before the admission to our ICU
* Known or suspected underlying immune deficiency (history of solid organ or stem cell transplantation, infection with human immunodeficiency virus, haematological malignancy, use of immunosuppressive medication (more than 0.1 mg /kg prednisone for >3 months, more than 1 mg/kg/day prednisone for >3 weeks or equivalent), chemotherapy/ radiotherapy in the year before ICU admission and any known humeral or cellular immune deficiency.
* Pregnancy
* Patient who do not consent for study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult ICU patients requiring prolonged mechanically ventilation (at least 7 days of supportive ventilation) and the presence of CMV seropositivity (Anti CMV IgG antibodies) will be screened for the possible inclusion.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The prevalence of cytomegalovirus reactivation in ICU patients requiring prolong mechanical ventilation | Till 4 weeks after the initiation of mechanical ventilation
  Percentage of total included patients (CMV seropositive IgG) who had viral load >1000/cc will be calculated.
The correlation of CMV viral load with the severity of illness . | Till 3 weeks after the cytomegalovirus reactivation
  Patients who had cytomegalovirus reactivation, the correlation will be explored between cytomegalovirus viral load with the severity of illness (total SOFA score).

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS)
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided